CLINICAL TRIAL: NCT01212302
Title: Optimizing Therapy With Aspirin and Clopidogrel. The BOchum CLopidogrel and Aspirin Plan to Improve Dual Antiplatelet Therapy.
Brief Title: Optimizing Aspirin and Clopidogrel Therapy (BOchum CLopidogrel and Aspirin Plan)
Acronym: BOCLAplan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Horst Neubauer, MD, Ruhr-University Bochum
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BOCLAplan01; F654R (Registry Identifier: F654R Ruhr-University Bochum)
Record Dates: First submitted 2010-09-29; First posted 2010-09-30 (Estimated); Results first posted 2011-09-16 (Estimated); Last update posted 2011-09-16 (Estimated); Status verified 2010-09

CONDITIONS: Coronary Artery Disease
Keywords: Clopidogrel; ASA; Low Response; Resistance
MeSH Terms: conditions — Coronary Artery Disease | interventions — Aspirin; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- aspirin, clopidogrel (Experimental): If the treatment with aspirin and/or clopidogrel is insufficient (platelet function testing) the dose was increased or the drug was changed (clopidogrel to ticlopidine or prasugrel)
  Interventions: Drug: Optimizing ASA and clopidogrel treatment

INTERVENTIONS:
Drug: Optimizing ASA and clopidogrel treatment — ASA 100 mg, ASA 300 mg, ASA 500 mg
  Clopidogrel 75 mg, Clopidogrel 150 mg, Ticlopidine 2x 250 mg, Prasugrel 10 mg. Intervention List:
  In the case of clopidogrel low-response, the maintenance dose was doubled (repeated loading dose followed by 150 mg daily), and when still ineffective ticlopidine or prasugrel, if available and not contraindicated, were used. ASA low-responders were treated by increasing the dose to 300 mg in a first step or to 500 mg ASA when the first modification was not sufficient.
  Other Names: ASA (aspirin), Clopidogrel (Plavix)

SUMMARY:
Dual antiplatelet therapy with acetylsalicylic acid (ASA, aspirin) and clopidogrel is of great importance for treatment following coronary stenting. Unfortunately the variable platelet inhibitory effectiveness compromises the antithrombotic benefit of dual antiplatelet therapy. The aim of this prospective single centre study was to reduce the low response incidence of dual antiplatelet therapy with ASA and clopidogrel based on a standardized therapy algorithm.

DETAILED DESCRIPTION:
Platelet function testing using whole blood aggregometry was performed 48 hours following coronary stenting (either acute coronary syndromes or stable coronary artery disease). The antiplatelet therapy included a loading dose of 600 mg clopidogrel and 500 mg ASA, followed by 75 mg clopidogrel and 100 mg ASA once daily. Clopidogrel low-response (CLR) and/or ASA (ASA low response) were treated according to a structured therapy plan.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stable coronary artery disease (CAD) or acute coronary syndromes (ACS) following percutaneous coronary intervention (PCI)

Exclusion Criteria:

* abnormal platelet count in patients,
* severe liver disorders,
* current gastrointestinal disorders,
* current infections,
* congestive heart failure,
* known bleeding disorders,
* treatment with bivalirudin or glycoprotein IIb/IIIa antagonists within the last 7 days.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2008-10; Primary Completion 2010-03 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Horst Neubauer, MD, Principal Investigator — Ruhr-University Bochum, Cardiovascular Center
Locations (1):
- Cardiovascular Center, Ruhr University Bochum, St. Josef - Hospital, Gudrunstrasse 56, Bochum, North Rhine-Westphalia, Germany

REFERENCES:
- [Background] Geisler T, Gawaz M, Steinhubl SR, Bhatt DL, Storey RF, Flather M. Current strategies in antiplatelet therapy--does identification of risk and adjustment of therapy contribute to more effective, personalized medicine in cardiovascular disease? Pharmacol Ther. 2010 Aug;127(2):95-107. doi: 10.1016/j.pharmthera.2010.04.017. Epub 2010 Jun 1. PMID 20570595
- [Background] Collet JP, Silvain J, Landivier A, Tanguy ML, Cayla G, Bellemain A, Vignolles N, Gallier S, Beygui F, Pena A, Montalescot G. Dose effect of clopidogrel reloading in patients already on 75-mg maintenance dose: the Reload with Clopidogrel Before Coronary Angioplasty in Subjects Treated Long Term with Dual Antiplatelet Therapy (RELOAD) study. Circulation. 2008 Sep 16;118(12):1225-33. doi: 10.1161/CIRCULATIONAHA.108.776757. Epub 2008 Sep 2. PMID 18765393
- [Background] Bonello L, Armero S, Ait Mokhtar O, Mancini J, Aldebert P, Saut N, Bonello N, Barragan P, Arques S, Giacomoni MP, Bonello-Burignat C, Bartholomei MN, Dignat-George F, Camoin-Jau L, Paganelli F. Clopidogrel loading dose adjustment according to platelet reactivity monitoring in patients carrying the 2C19*2 loss of function polymorphism. J Am Coll Cardiol. 2010 Nov 9;56(20):1630-6. doi: 10.1016/j.jacc.2010.07.004. Epub 2010 Aug 12. PMID 20708365
- [Background] Neubauer H, Lask S, Engelhardt A, Mugge A. How to optimise clopidogrel therapy? Reducing the low-response incidence by aggregometry-guided therapy modification. Thromb Haemost. 2008 Feb;99(2):357-62. doi: 10.1160/TH07-10-0624. PMID 18278186
- [Background] Angiolillo DJ, Shoemaker SB, Desai B, Yuan H, Charlton RK, Bernardo E, Zenni MM, Guzman LA, Bass TA, Costa MA. Randomized comparison of a high clopidogrel maintenance dose in patients with diabetes mellitus and coronary artery disease: results of the Optimizing Antiplatelet Therapy in Diabetes Mellitus (OPTIMUS) study. Circulation. 2007 Feb 13;115(6):708-16. doi: 10.1161/CIRCULATIONAHA.106.667741. Epub 2007 Jan 29. PMID 17261652
- [Derived] Neubauer H, Kaiser AF, Endres HG, Kruger JC, Engelhardt A, Lask S, Pepinghege F, Kusber A, Mugge A. Tailored antiplatelet therapy can overcome clopidogrel and aspirin resistance--the BOchum CLopidogrel and Aspirin Plan (BOCLA-Plan) to improve antiplatelet therapy. BMC Med. 2011 Jan 12;9:3. doi: 10.1186/1741-7015-9-3. PMID 21226927

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Medical Clinic, 504 patients 2007-2010
Pre-assignment Details: post coronary stenting
Period: Overall Study
Arm/Group | Aspirin, Clopidogrel
Started | 504
Completed | 504
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Aspirin, Clopidogrel
Number analyzed (Participants) | 504
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 294
  >=65 years | 210
Age Continuous [Mean (Standard Deviation); unit: years] | 64.3 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 154
  Male | 350
Region of Enrollment [Number; unit: participants]
  Germany | 504

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Were Responders or Low-Responders of Antiplatelet Therapy as a Result of Whole Blood Aggregometry Testing (See Outcome Measure Description)
Description: In patients treated with aspirin and clopidogrel aggregometry was performed and depending on the results the patients were either responder or low-responder of antiplatelet therapy.
  The following definitions were used for clopidogrel low response (CLR: >5 ohm when stimulated with adenosine diphosphate (ADP) 5 μM) and ASA low response (ALR: >0 ohm;stimulated with arachidonic acid 10 μM) with the ChronoLog 590 aggregometer. In the case of low-response alternative antiplatelet therapy was modified according to the study plan (see protocol section).
Time Frame: 2 years
Population: Sample size calculation: With the assumption that the incidence of clopidogrel low response was at least 20% and ASA low response 10%. Choosing a power of 97.5% and a two-sided value of 0.05, an overall sample size was required of at least 400 patients. To compensate for a possible loss of follow-up, we aimed for inclusion of approx. 500 patients.
Measure: Number (95% Confidence Interval); unit: participants
Groups:
- Clopidogrel Low Response: If the treatment with aspirin and/or clopidogrel is insufficient (platelet function testing) the dose was increased or the drug was changed (clopidogrel to ticlopidine or prasugrel)
Arm/Group | Clopidogrel Low Response
Number analyzed (Participants) | 504
participants | 155 [155 to 155]

ADVERSE EVENTS:
Arm/Group | Aspirin, Clopidogrel
Serious Adverse Events (participants affected / at risk) | 0/504
Other Adverse Events (participants affected / at risk) | 0/504

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No